CLINICAL TRIAL: NCT02760459
Title: Effects of Perioperative Intravenous Dexamethasone on the Severity of Persistent Postsurgical Pain After Total Knee Arthroplasty : A Prospective, Randomized, Double-blind, Placebo-controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Nitchanant Kitcharanant, MD, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORT-2558-03245; 054/2559 (Other Grant/Funding Number: Faculty of medicine, Chiangmai university fund)
Record Dates: First submitted 2016-05-01; First posted 2016-05-03 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dexamethasone (Active Comparator): The steroid group will receive Dexamethasone 10 mg IV immediately prior to induction of spinal anesthesia and will receive a second and third dose of Dexamethasone 10 mg IV postoperatively at 24 and 48 hrs.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): The control group will receive sterile normal saline solution, serving as placebo, IV immediately prior to induction of spinal anesthesia and will receive a second and third dose of placebo IV postoperatively 24 and 48 hrs. Both Dexamethasone and normal saline solution will be administered as an IV push.
  Interventions: Drug: Normal saline solution

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Dexamethasone
Drug: Normal saline solution
  Arms: Placebo

SUMMARY:
To compare the effects of perioperative intravenous Dexamethasone with a placebo on the severity of persistent postsurgical pain after total knee arthroplasty.

DETAILED DESCRIPTION:
It is not clear whether perioperative intravenous Dexamethasone has an effect on severity of persistent postsurgical pain (PPSP) after total knee arthroplasty (TKA). The research hypothesis is that TKA patients experience less severe PPSP after administration of perioperative intravenous Dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years (45)
* Primary knee osteoarthritis diagnosed using the American College of Rheumatology criteria (46)
* Undergoing elective, primary and unilateral total knee arthroplasty
* American Society of Anesthesiology (ASA) physical status class 1-3
* BMI < 40 kg/m2

Exclusion Criteria:

* History of active rheumatic diseases
* History of previous musculoskeletal injury of the same knee for excluding patients with secondary knee osteoarthritis
* History of previous surgery on the same knee
* History of adverse effects from medications to be used in this study
* Contraindication to spinal anesthesia
* History of psychiatric disorders or cognitive impairment
* Contraindication to corticosteroid agents
* Poorly controlled diabetes mellitus (HbA1C > 7.5)
* Poorly controlled hypertension
* History of ischemic heart disease or peripheral arterial disease or cerebrovascular disease
* Hepatic insufficiency (Child-Pugh score > 5)
* Renal insufficiency (Creatinine clearance < 30 mL/min)
* History of cataracts or glaucoma or ocular hypertension
* History of steroid or immunosuppressive drug use within 6 months of surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Modified WOMAC scores for pain at 12 weeks postoperative | 12 weeks
  using the modified Thai version of the Western Ontario and McMaster (WOMAC) osteoarthritis index for knee osteoarthritis questionnaire

SECONDARY OUTCOMES:
Visual analogue scales for pain during a five-meter walk (0-100) | postoperatively at 24, 30, 48, 54, 72 hrs
Visual analogue scales for pain during 45 degree active knee flexion (0-100) | postoperatively at 6, 24, 30, 48, 54, 72 hrs
Visual analogue scales for current pain at rest in a supine position (0-100) | postoperatively at 6, 24, 30, 48, 54, 72 hrs
Visual analogue scales for maximum pain at rest over the last 24 hours and minimum pain at rest over the last 24 hours (0-100) | postoperatively at 0-24, 24-48, 48-72 hrs
Visual analogue scale values for nausea (0-100) | postoperatively at 6, 24, 30, 48, 54, 72 hrs
Opioid consumption (mg.) | during the first 0-24, 24-48, and 48-72 hrs
Anti-emetic medicine consumption (mg.) | during the first 0-24, 24-48, and 48-72 hrs
Maximum degree of active knee flexion | postoperatively at 24, 48, 72 hrs, 2 weeks, 6 weeks, and 12 weeks
Modified WOMAC scores for pain | postoperatively at weeks 2 and 6
  using the modified Thai version of the Western Ontario and McMaster (WOMAC) osteoarthritis index for knee osteoarthritis questionnaire
Wound complications | evaluated postoperatively at weeks 2, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Nitchanant Kitcharanant, MD, Principal Investigator — Department of Orthopedics, Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Orthopedics, Chiang Mai University, Chiang Mai, ChiangMai, Thailand

REFERENCES:
- [Background] 1. Callahan CM, Drake BG, Heck DA, Dittus RS. Patient outcomes following tricompartmental total knee replacement. A meta-analysis. JAMA. 1994;271(17):1349-57. 2. Grosu I, Lavand'homme P, Thienpont E. Pain after knee arthroplasty: an unresolved issue. Knee Surg Sports Traumatol Arthrosc. 2014;22(8):1744-58.
- [Derived] Kitcharanant N, Leurcharusmee P, Atthakomol P, Jingjit W. Perioperative intravenous dexamethasone did not reduce the severity of persistent postsurgical pain after total knee arthroplasty: a prospective, randomized, double-blind, placebo-controlled trial. J Orthop Surg Res. 2024 Dec 19;19(1):854. doi: 10.1186/s13018-024-05362-y. PMID 39702151